CLINICAL TRIAL: NCT05107193
Title: Assessment of Prospective Real-world Outcomes Based on Single-patient Protocol Data Collection of Afatinib (GILOTRIF®) Use in Patients With Solid Tumors Harboring NRG1 Gene Fusions
Brief Title: Afatinib (GILOTRIF®) in Patients Suffering From Tumors Harboring Neuregulin 1 (NRG1) Gene Alterations (Specifically NRG1 Gene Fusion-positive Advanced Solid Tumors)
Status: No longer available | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0344
Record Dates: First submitted 2021-09-16; First posted 2021-11-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumors
Keywords: NRG1 fusion
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: afatinib — afatinib
  Other Names: GILOTRIF®

SUMMARY:
Gene fusions are defined as two separate genes joined together (gene 1, gene 2), generating a novel fusion gene. NRG1 fusions are rare and complex with regard to the fusion/fusion partner. The specific NRG1 gene fusion will be identified by a specialized molecular testing lab.

DETAILED DESCRIPTION:
Afatinib is provided on a single-patient protocol basis to patients suffering from tumors harboring NRG1 fusions, a disease for which no satisfactory authorised alternative therapy exists.

In the context of this mechanism it is planned to collect and analyze limited clinical data in order to investigate the safety and efficacy of afatinib in patients with advanced and/or metastatic solid tumours harboring NRG1 gene fusions.

ELIGIBILITY:
Inclusion Criteria to participate in this program:

* Confirmed diagnosis of an advanced, unresectable and/or metastatic tumor harboring NRG1 gene fusions characterized as follows:

  * Gene 1: NRG1 (prerequisite: conservation of the epidermal growth factor (EGF) domain - this will be identified by the lab performing the molecular testing)
  * Gene 2: All fusion partners are allowed (prerequisite: the region must be a coding region - this will be identified by the lab performing the molecular testing)
* Patient must have measurable or evaluable lesions (according to RECIST 1.1).
* At least 18 years of age at the time of consent.

Exclusion Criteria:

* Treatment with a systemic anti-cancer therapy or investigational drug within 14 days or 5 half-lives (whichever is shorter) of the first treatment with the study medication.
* Tumors carrying additional gene mutations other than NRG1 fusion where FDA-approved targeted therapy is available
* Prior treatment with a therapy targeting erythroblastic leukemia viral oncogene homologue receptors (ErbB)
* Any patient considered ineligible by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com